CLINICAL TRIAL: NCT02095314
Title: Antibody Persistence After Primary Doses, Immune Response and Safety After Doses of Pentabio Vaccine in Indonesian Children at 18-24 Months of Age
Brief Title: Antibody Persistence, Immune Response and Safety After Doses of Pentabio Vaccine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Booster Penta 0413
Record Dates: First submitted 2014-03-19; First posted 2014-03-24 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: DTP-HB-Hib; Pentavalen; Pentabio; Booster

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pentavalen (Experimental): Pentabio Vaccine One dose corresponds to 0.5ml The vaccine shall be given intramuscularly
  Interventions: Biological: Pentavalen

INTERVENTIONS:
Biological: Pentavalen — Batch 5010613
  Other Names: Pentabio vaccine; DPT-HB-Hib

SUMMARY:
Measure antibody persistence prior to booster administration of Pentabio vaccine.

DETAILED DESCRIPTION:
Number and percentage of children with anti diphtheria, titer and anti tetanus titer >= 0.01 IU/ml, anti HBs >=10mIU/ml, anti Hib >=0.15ug/ml prior to booster administration.

ELIGIBILITY:
Inclusion Criteria:

* Children, 18-24 months of age
* Subjects who had completed the primary series of Pentabio vaccine in the previous trial
* Father, mother, or legally acceptable representative have been informed properly regarding the study and signed the informed consent form
* Subject's parents commit to comply with the instruction

Exclusion Criteria:

* Subjects concomitantly enrolled or scheduled to be enrolled in another trial
* Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature >=37.5oC on Day 0)
* Known history of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
* Known history of allergy to any component of the vaccines (e.f. formaldehyde)
* Known history of acquired immunodeficiency (including HIV infection)
* Subject who has received a treatment likely to alter immune response in the previous 4 weeks (e.g intravenous immunoglobulin, blood-derived products or long term corticotherapy (>2 weeks)
* Subject receives other vaccination within 1 month prior to inclusion
* Any abnormality or chronic disease justified by investigator that might interfere assessment of the trial objectives
* Infant with a known history of diphtheria, tetanus, pertussis, Hepatitis B and Hib infection

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 399 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Geomoteric mean titer prior to booster administration of Pentabio vaccine | visit 1
  The number and percentage of children with anti diphtheria titer and anti tetanus titer >=0.01 IU/ml anti HBs >=10 mIU/ml, anti Hib >=0.15 ug/ml prior to booster administration.

SECONDARY OUTCOMES:
Protectivity of Pentabio vaccine 1 month after the booster dose | 1 month
  Serological response to diphtheria, tetanus, pertussis and Hib (Geometric Mean Titer)
Serological response to diphtheria, tetanus, pertussis, hepatitis B and PRP-T before and 1 month after the booster dose | 1 month
  Geometric mean titer to diphtheria, tetanus, pertussis, Hepatitis B and Hib before immunization and 1 month after immunization
Seroconversion and seroprotection before and 1 month after the booster dose | 1 month
  The changes of serological response before and after booster dose
Number of participants with adverse events | 1 month
  Local and systemic reaction within 28 days after immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Kusnandi Rusmil, MD, Principal Investigator — Department of Child Health, School of Medicine Padjadjaran University; Hartono Gunardi, MD, Principal Investigator — Department of Child Health, School of Medicine, University of Indonesia
Locations (6):
- Indonesia (6):
  - Jatinegara Primary Health Center, Jakarta, Jakarta Special Capital Region
  - Mampang Prapatan Primary Health Center, Jakarta, Jakarta Special Capital Region
  - Tebet Primary Health Center, Jakarta, Jakarta Special Capital Region
  - Garuda Primary Health Center, Bandung, West Java
  - Ibrahim Adjie Primary Health Center, Bandung, West Java
  - Puter Primary Health Centre, Bandung, West Java

REFERENCES:
- [Derived] Gunardi H, Rusmil K, Fadlyana E, Soedjatmiko, Dhamayanti M, Sekartini R, Tarigan R, Satari HI, Medise BE, Sari RM, Bachtiar NS, Kartasasmita CB, Hadinegoro SRS. DTwP-HB-Hib: antibody persistence after a primary series, immune response and safety after a booster dose in children 18-24 months old. BMC Pediatr. 2018 May 28;18(1):177. doi: 10.1186/s12887-018-1143-6. PMID 29804542